CLINICAL TRIAL: NCT01858844
Title: EVALUATION OF THE EFFECTS OF MANUAL CHEST COMPRESSION TECHNIQUE IN INFANTS WITH PULMONARY ATELECTASIS- Clinical CONTROLLED TRIAL
Brief Title: Chest Compression Technique in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, PhD, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEST COMPRESSION TECHNIQUE
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHEST COMPRESSION TECHNIQUE 2 (Active Comparator): The CCT was held only once. Prior to the start of data collection the patients were placed in supine position, with the slope of the headboard of the bed in 30 degrees for collection of signs of respiratory distress (runs), RR(respiratory rate)(timer for 1 minute); HR (heart rate) and SpO2(oxygen saturation) through pulse oximetry in infants without atelectasis.
  Interventions: Other: CHEST COMPRESSION TECHNIQUE (CCT)
- CHEST COMPRESSION TECHNIQUE (Experimental): The CCT was held only once. Prior to the start of data collection the patients were placed in supine position, with the slope of the headboard of the bed in 30 degrees for collection of signs of respiratory distress (runs), RR (timer for 1 minute); HR and SpO2 through pulse oximetry in infants with atelectasis.
  Interventions: Other: CHEST COMPRESSION TECHNIQUE (CCT)

INTERVENTIONS:
Other: CHEST COMPRESSION TECHNIQUE (CCT) — The CCT was held with the placement of one of the hands were not engaged in. The following has been applied a symmetric oblique direction, pressure from top to bottom on the half thorax rib cage so that it went according to the complacency of the ribcage. This pressure was applied in the expiratory phase and held for 10 seconds, totaling 6 repetitions of the maneuver during 60 seconds. The other hand held on the contralateral iliac crest to stabilize the patient. The technique was held during 5 consecutive minutes with range of a respiratory incursion every 60 seconds. Immediately after and 10 minutes after the end of the application of the technique, the data was measured again.

SUMMARY:
Evaluate the effect of chest manual compression technique (CCT) in the variables of oxygenation, hemodynamic and respiratory work in infants with respiratory diseases that are associated with atelectasis.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Infants (29 days to 24 months of age).
* After the legal representatives of the patients have read agreed and signed an informed consent
* Infants diagnosed with atelectasis by medical staff, with chest x-ray with opacification directors
* Respiratory disease

Group B (control group)

* Infants whose inpatient diagnosis has not been respiratory ailments that did not show any pain at the time of the evaluation.

For the control group followed the same evaluation criteria of group A.

Exclusion Criteria:

* Infants with respiratory disorders that don't have with atelectasis
* Infants who showed signs of irritability or intense crying at the time of evaluation

Ages: 29 Days to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in clinical signs | baseline, within one minute after and 10 min after CCT
  Variation in clinical signs of oxygenation and respiratory and cardiac frequency

SECONDARY OUTCOMES:
Changes in signs of respiratory distress | baseline, within one minute after and 10 min after CCT
  Signs of respiratory distress

CONTACTS AND LOCATIONS:
Overall Officials: Evelim Leal de Freitas D Gomes, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Hospital do Mandaqui, São Paulo, São Paulo, Brazil